CLINICAL TRIAL: NCT04464122
Title: Rediscovering Biomarkers for the Diagnosis and Early Treatment Response in NEN. REBORN Study
Brief Title: Rediscovering Biomarkers for the Diagnosis and Early Treatment Response in NEN (REBORN)
Acronym: REBORN
Status: Recruiting | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea M. Isidori, Full Professor, University of Roma La Sapienza
Other Study IDs: Reborn Study
Record Dates: First submitted 2020-07-03; First posted 2020-07-09 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Neuroendocrine Tumors; Neuroendocrine Neoplasm; Neuroendocrine Tumor Grade 1; Neuroendocrine Tumor Grade 2; Neuroendocrine Carcinoma
Keywords: Neuroendocrine Tumours; Prognostic markers; Tumour educated platelets; angiogenesis; immune function
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoma, Neuroendocrine | interventions — Somatostatin; Drug Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Neuroendocrine toumor group: 30 patients (18-80 years, males and females) affected by histologically-proven neuroendocrine neoplasms, locally advanced or metastatic, originating from pulmonary or gastro-entero-pancreatic (GEP) tract, candidate to medical therapy.
  Interventions: Drug: Somatostatin analog; chemotherapy
- Control group: Patients affected by other non-malignant endocrine disease, e.g. benign thyroid disfunction (18-80 years, males and females)

INTERVENTIONS:
Drug: Somatostatin analog; chemotherapy — According to current ENETS guidelines, patients will be treated by somatostatin analogs or chemotherapy, recommended respectively as first line therapy in neuroendocrine tumours or neuroendocrine neoplasms.
  Groups: Neuroendocrine toumor group

SUMMARY:
This is a multicentre, controlled, observational prospective study on new biomarkers, as immune profiling, angiogenetic markers and circRNA from TEPs in the diagnosis and in the evaluation of treatment response in pulmonary and gastro-entero-pancreatic NENs.

DETAILED DESCRIPTION:
Neuroendocrine Neoplasm (NEN) are heterogeneous disease in terms of origin, localization and clinical presentation. Annual incidence of NEN is increasing in the last 30 years, even if the reasons underlying this rise have not been completely identified.

Many biomarkers have been used in the diagnosis and follow-up of patients with NEN. In non-functioning NEN general tumor markers, such as chromogranin A (CgA) and neuron specific enolase (NSE), are commonly used but their sensibility and specificity are quite low.

Recently, high-throughput tissue microarray and immunohistochemistry assessments have been performed to observe the expression pattern of new potential markers for NEN. In order to overcome limitations of tissue acquisition, the use of liquid biopsies has been advocated. It has been reported that tumor-educated platelets (TEPs) may easily enable blood-based cancer diagnostics. TEPs take up tumor-derived secreted membrane vesicles containing RNAs, of which circular RNAs (circRNAs) that can serve as a potential biomarker source for cancer diagnostics. This innovative approach in cancer detection has not yet been transferred to the NEN field.

Flow cytometric analysis furnishes important insights into the immune status by providing information about the numbers and phenotypes of the immune cells, which are known to be altered in many types of neoplasms. In NEN, leukocytes subpopulations and peripheral blood mononuclear cells (PBMCs) are not been completely investigated but immunological alterations could represent a signal of neoplastic spread.

Inflammatory and angiogenetic pathways' involvement in NEN behavior has recently received increasing attention. It is well known that NEN are known to be highly vascularized neoplasms and somatostatin analogues (SSA), used as first line drugs for most well differentiated NEN, can reduce tumour proliferation by various direct and indirect mechanism including the inhibition of angiogenesis.

Tumor angiogenesis is a complicated process consisting of several steps, the angiogenesis cascade, regulated by endogenous and exogenous factors, including the system Angiopoietin-1 (Ang-1) and -2 (Ang-2) / Tie2 and Prokineticins. These systems are involved in neoplastic angiogenesis and inflammation in various types of cancer. Despite these evidences, the role of inflammatory and angiogenic factors in NEN detection and follow-up has not been completely clarified.

The aim of the study is to evaluate immune profiling, angiogenetic markers and circularRNA sequencing in patients affected by locally advanced or metastatic pulmonary or GEP NENs and controls. Moreover, NENs patients will be evaluated also after 1 and 3 months of first line medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven NENs, locally advanced or metastatic, originating from pulmonary or gastro-entero-pancreatic (GEP) tract, candidate to first line medical therapy (study group);
* Patients affected by other non-malignant endocrine disease, e.g. benign thyroid disfunction (control group).

Exclusion Criteria:

* Severe chronic kidney disease (stage 4-5);
* Clinical or laboratory signs of significant respiratory, cardiological and hepatobiliary disease;
* Other non-neuroendocrine malignancies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically-proven NENs, locally advanced or metastatic, originating from pulmonary or gastro-entero-pancreatic tract
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2025-09-14 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the modification of the angiogenetic mediator sTie2 after treatment. | baseline - + 1 month - +3 months
  Modification of sTie (soluble Tie2) after treatment

SECONDARY OUTCOMES:
To evaluate the difference in the angiogenetic mediator sTie2 between patients and controls | baseline
  Comparison of basal levels of sTie between patients and controls
To validate the use of circular RNAs from TEPs in NEN diagnosis | baseline
  Validation of the use of circular RNAs sequencing from tumor educated platelets (TEPs) in NETs diagnosis, through the comparison between patients and controls
To evaluate the changing in circular RNAs from TEPs in NEN patients after somatostatin analogs treatment | baseline - + 1 month - +3 months
  Modification in circular RNAs sequencing from tumor educated platelets (TEPs) in patients after treatment
To compare circular and cellular angiogenesis mediators between patients and controls | baseline
  Comparison of basal level of other circular and cellular angiogenesis mediators between patients and controls (Angiogenic factors: ANG1, ANG2, FGF1, FGF2, NRP1, NRP2, VEGFA, VEGFB, VEGFC, HIF1A, NOS3, PROK1, PROK2; Cytokines: CCL11, CCL2, CXCL1, CXCL10, CXCL5, CXCL6, CXCL9, IL1B, IL6, TNF; Receptors and other angiogenic factors: VEGFR1, VEGFR2, TIE2, PDGFR, TGFBR, MMP14, MMP2, MMp9, TIMP1, TIMP2, TIMP3, PROKR1, PROKR2)
To evaluate the changing in circular and cellular angiogenesis mediators after treatment. | baseline - + 1 month - +3 months
  Modification of other circular and cellular angiogenesis mediators in patients after treatment (Angiogenic factors: ANG1, ANG2, FGF1, FGF2, NRP1, NRP2, VEGFA, VEGFB, VEGFC, HIF1A, NOS3, PROK1, PROK2; Cytokines: CCL11, CCL2, CXCL1, CXCL10, CXCL5, CXCL6, CXCL9, IL1B, IL6, TNF; Receptors and other angiogenic factors: VEGFR1, VEGFR2, TIE2, PDGFR, TGFBR, MMP14, MMP2, MMp9, TIMP1, TIMP2, TIMP3, PROKR1, PROKR2)
To quantify PBMC subpopulation in patients and controls | baseline
  Quatification of peripheral blood mononuclear cells (PBMC) subpopulations in patients and controls
To evaluate the modification of PBMC subpopulation in patients after treatment | baseline - + 1 month - +3 months
  Modification of peripheral blood mononuclear cells (PBMC) subpopulations in patients after treatment
To compare classical neuroendocrine markers serum levels between patients and controls | baseline
  Comparison of basal serum level of classical neuroendocrine markers (chromogranin a and neuron specific enolase) between patients and controls
To evaluate the modification of classical neuroendocrine markers in patients after treatment | baseline - + 1 month - +3 months
  Modification of classical neuroendocrine markers (chromogranin a and neuron specific enolase) in patients after treatment
To evaluate infectious diseases frequency and severity between patients and controls | baseline
  Frequencies and severity of infectious diseases will be evaluated by modified Infectious Diseases Questionnaire (GNC). This questionnaire includes questions on infectious diseases of upper and lower respiratory tract, gastrointestinal tract, skin and urogenital tract contracted during the previous 12 months. Questions investigate on the number and duration of infections, necessity of antibiotic or antifungal therapy, hospital stay and days of absence from work. Final score represents the frequency of infections. Moreover, some questions investigate possible susceptible or protective factors for infectious diseases: vaccinations, use of corticosteroids, concomitant diseases, previous appendectomy, tonsillectomy, adenoidectomy, splenectomy or thymectomy.
To evaluate the difference in quality of life questionnaire in patients and controls | baseline
  Quality of life will be evaluated by the Physical Component score and the Mental Component score of the self-administered questionnaire SF-36-Item Health Survey questionnaire. This questionnaire measures eight scales: physical functioning, role physical, bodily pain, general health (physical component) and vitality, social functioning, role emotional, mental health (mental component).
  Interpretation of the score will be the following: at each item of the questionnaire corresponds a percentage value (from 0% to 100%). The average of the single items constitutes the scale total percentage (from 0% to 100%); missing data are not considered during calculation. High score defines a more favorable health state.
To evaluate the modification in quality of life questionnaire in patients after treatment | baseline - + 1 month - +3 months
  Quality of life will be evaluated by the Physical Component score and the Mental Component score of the self-administered questionnaire SF-36-Item Health Survey questionnaire. This questionnaire measures eight scales: physical functioning, role physical, bodily pain, general health (physical component) and vitality, social functioning, role emotional, mental health (mental component).
  Interpretation of the score will be the following: at each item of the questionnaire corresponds a percentage value (from 0% to 100%). The average of the single items constitutes the scale total percentage (from 0% to 100%); missing data are not considered during calculation. High score defines a more favorable health state.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Isidori, MD, PhD, Principal Investigator — Department of Experimental Medicine, Sapienza University of Rome
Locations (1):
- Andrea M Isidori, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sol N, Wurdinger T. Platelet RNA signatures for the detection of cancer. Cancer Metastasis Rev. 2017 Jun;36(2):263-272. doi: 10.1007/s10555-017-9674-0. PMID 28681241
- [Background] Joosse SA, Pantel K. Tumor-Educated Platelets as Liquid Biopsy in Cancer Patients. Cancer Cell. 2015 Nov 9;28(5):552-554. doi: 10.1016/j.ccell.2015.10.007. PMID 26555171
- [Background] Fiedler U, Augustin HG. Angiopoietins: a link between angiogenesis and inflammation. Trends Immunol. 2006 Dec;27(12):552-8. doi: 10.1016/j.it.2006.10.004. Epub 2006 Oct 12. PMID 17045842
- [Background] Monnier J, Samson M. Prokineticins in angiogenesis and cancer. Cancer Lett. 2010 Oct 28;296(2):144-9. doi: 10.1016/j.canlet.2010.06.011. Epub 2010 Jul 14. PMID 20633984
- [Background] Best MG, Sol N, Kooi I, Tannous J, Westerman BA, Rustenburg F, Schellen P, Verschueren H, Post E, Koster J, Ylstra B, Ameziane N, Dorsman J, Smit EF, Verheul HM, Noske DP, Reijneveld JC, Nilsson RJA, Tannous BA, Wesseling P, Wurdinger T. RNA-Seq of Tumor-Educated Platelets Enables Blood-Based Pan-Cancer, Multiclass, and Molecular Pathway Cancer Diagnostics. Cancer Cell. 2015 Nov 9;28(5):666-676. doi: 10.1016/j.ccell.2015.09.018. Epub 2015 Oct 29. PMID 26525104
- [Background] Harris AL, Reusch P, Barleon B, Hang C, Dobbs N, Marme D. Soluble Tie2 and Flt1 extracellular domains in serum of patients with renal cancer and response to antiangiogenic therapy. Clin Cancer Res. 2001 Jul;7(7):1992-7. PMID 11448916